CLINICAL TRIAL: NCT02090231
Title: Phase 2 Study of rTMS on Poststroke Dysphagia
Brief Title: The Effect of Repetitive Transcranial Magnetic Stimulation for Poststroke Dysphagia Recovery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, vghtpe user, Po-Yi Tsai, MD, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-10-022OB
Record Dates: First submitted 2014-03-11; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Stroke; Dysphagia
Keywords: stroke; dysphagia; rTMS
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real 5 Hz rTMS (Experimental): real 5 Hz rTMS, 10 minutes per day, for 10 weekdays.
  Interventions: Device: rTMS, Magstim Rapid2
- sham 5 Hz rTMS (Sham Comparator): sham 5Hz rTMS, 10 minutes per day, for 10 weekdays.
  Interventions: Device: rTMS, Magstim Rapid2

INTERVENTIONS:
Device: rTMS, Magstim Rapid2 — 5 Hz rTMS

SUMMARY:
Dysphagia is one of severe complications among stroke survivors. Dysphagia is usually associated with high levels of morbidity, mortality, and financial cost. In recent years, repetitive transcranial magnetic stimulation (rTMS) has shown promise to facilitate poststroke dysphagia. However, most researches were preliminary studies in the past. The present study aims to investigate the immediate and long-term efficacy of high frequency rTMS on chronic dysphagic patients.

DETAILED DESCRIPTION:
rTMS protocol: 5 Hz real or sham stimulation, 10 minutes per day, for 10 week-days.

ELIGIBILITY:
Inclusion Criteria:

* Poststroke dysphagia more than 3 months

Exclusion Criteria:

* Hx of seizure or a metalic device in brain or chest

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-07 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Dysphagia severity on Aus TOMs swallowing score | up to 3 months

SECONDARY OUTCOMES:
Imaging evidence with video-esophagography | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Tsui-Fen Yang, MD, Principal Investigator — No. 201, Shih- Pai Rd, Sec. 2, Taipei, 11217 Taiwan.
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan